CLINICAL TRIAL: NCT07025993
Title: Effects of Muscle Energy Technique Versus Cervical and Scapulothoracic Stabilization Exercises on Pain, Disability and Craniovertebral Angle in Patients With Upper Crossed Syndrome
Brief Title: Effects of Muscle Energy Technique Versus Cervical and Scapulothoracic Stabilization Exercises in Upper Crossed Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jaazba- REC/RCR&AHS 24/0137
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Upper Cross Syndrome
Keywords: Posture; Neck Pain; Upper Cross Syndrome; Exercise
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Other: Muscle Energy Technique
- Group B (Experimental)
  Interventions: Other: Eccentric muscle energy technique

INTERVENTIONS:
Other: Muscle Energy Technique — Eccentric muscle energy technique was applied to subjects' cervical spine. The cervical spine will brought to the barrier of motion in each plane i.e. flexion/extension, lateral bending and rotation. Then subjects will asked to push their heads into the direction opposite that of the barrier. The therapist provided isometric resistance for 3- 5 seconds, after which the subjects relaxed their muscles completely and the therapist applied stretch.
  Arms: Group A
Other: Eccentric muscle energy technique — Eccentric muscle energy technique was applied to subjects' cervical spine. The cervical spine will brought to the barrier of motion in each plane i.e. flexion/extension, lateral bending and rotation. Then subjects will asked to push their heads into the direction opposite that of the barrier. The therapist provided isometric resistance for 3- 5 seconds, after which the subjects relaxed their muscles completely and the therapist applied stretch. Three to five repetitions will performed.
  Arms: Group B

SUMMARY:
This study will be a randomized clinical trial and will be conducted in Younus Hospital, Tehsil headquarters hospital Daska, and Riphah Rehabilitation Clinic Lahore. Non-probability consecutive sampling will be used to collect the data. A sample size of 40 subjects with an age group between 18-65 years will be taken. Data will be collected from the patients having present complaints of Neck pain associated with upper cross syndrome. Outcome measures will be taken using the Numeric Rating Pain Scale (NRPS) for pain and the Neck disability index (NDI) for neck functional health and craniovertebral angle for posture. An informed consent will be taken. Subjects will be selected based on inclusion and exclusion criteria and will be equally divided into two groups by a random number generator table. Both Groups will receive Moist Hot Pack, Cervical segmental mobilizations, and Free Neck Exercises (AROMs), while Group A will receive Muscle energy technique(eccentric muscle energy technique for the cervical spine with Mets for upper trapezius, Suboccipitalis and pectoralis muscle), and Group B will receive cervical and scapulothoracic stabilization exercises(axial elongation exercise, craniocervical flexion, cervical extension and Cervico-scapulothoracic stabilization exercises). Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

DETAILED DESCRIPTION:
Neck pain is one of the most commonly occurring musculoskeletal disorders if left untreated can lead to severe complications. Cervical spine and soft tissue disorders e.g. muscles, ligaments, discs, facet joints, etc. are major causes of neck pain while neck pain caused by postural abnormality is termed as upper cross syndrome. Upper crossed syndrome (UCS) characterizes a prevalent postural dysfunction involving dysfunctional tone in the musculature of the neck, shoulders, and upper back that cross between the dorsal and the ventral sides of the body. This condition is given its name because an "X," in other words a cross, can be drawn across the upper body. One arm of the cross indicates the muscles that are typically tight/overly facilitated and the other arm of the cross indicates the muscles that are typically weak/overly inhibited. There are two types of muscles present in our body - the postural muscles such as pectoralis major, upper trapezius, and sternocleidomastoid, and other phasic muscles such as deep-neck flexors, and lower trapezius. In Upper Cross Syndrome (UCS) there is tightness of the upper trapezius and levator scapula on the dorsal side crosses with tightness of the pectoralis major and minor. Weakness of the deep cervical flexors, ventrally, crosses with weakness of the middle and lower trapezius. This pattern of imbalance creates joint dysfunction, particularly at the Atlanto-occipital joint, C4-C5 segment, cervicothoracic joint, glen humeral joint, and T4-T5 segment. Specific postural changes are seen in UCS, including forward head posture, increased cervical Lordosis and thoracic kyphosis, elevated and protracted shoulders, and rotation or abduction and winging of the scapulae. The main risk factor for developing UCS is maintaining an abnormal posture for a prolonged duration. Some daily activities that involve bad postures are often occupation-related. Repetitive tasks or continuous work for long hours can aggravate postural deviations. Because of increased work stress and a sedentary lifestyle, society is becoming more flexion-addicted attitude. In which people tend to frequently stoop forward. This is seen in office workers and students who tend to sit at a desk for prolonged periods, slouching forward to see the computer screen. Therefore, once muscle dysfunction starts, traditional muscle imbalance trends and altered posture follow. Head, neck structures can set limits on head's range of motion (ROM) and cause discomfort to the neck, mid-back muscle spasm/tightness, and decreased range of motion.

Understanding of which intervention yields better outcomes for pain relief, reduction in disability, and improvement in craniovertebral angle is crucial for optimizing treatment strategies for upper crossed syndrome patients. This study seeks to provide evidence-based guidance to clinicians regarding the most effective therapeutic approach. Considering the high prevalence of Upper Cross syndrome in the modern world, this study aims to check the effects of METs versus cervical and scapula-thoracic stabilization exercises on pain, disability and craniovertebral angle in patients with Upper Cross syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Both gender diagnosed with upper crossed syndrome
* Patient having neck pain of 4 to 12 weeks
* Pain reported on NRPS score ˃6/10 in the neck region
* Subjects agree to sign the written consent form.

Exclusion Criteria:

* Exclusion criteria Patients were excluded if they were diagnosed with the following conditions for ˃6 months
* Tuberculosis, carcinoma, heart disease, and osteoporosis
* Neural disorders due to prolapsed intervertebral disc
* Any trauma or localized infection in neck region
* Upper motor neuron disease, cervical stenosis, and metabolic diseases in bone and joint
* Hyper flexibility
* Open sores
* Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants
* Psychiatric diseases such as phobia/obsession and depression
* Allergy to hot pack

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Pain Scale (NRPS) | Baseline, 4th Week
  The patient's level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain".
Neck disability index (NDI) | Baseline, 4th Week
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain-related disability
Craniovertebral angle (CVA) | Baseline, 4th Week
  The craniovertebral angle is identified as the intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mujawar JC, Sagar JH. Prevalence of Upper Cross Syndrome in Laundry Workers. Indian J Occup Environ Med. 2019 Jan-Apr;23(1):54-56. doi: 10.4103/ijoem.IJOEM_169_18. PMID 31040591
- [Background] Chang MC, Choo YJ, Hong K, Boudier-Reveret M, Yang S. Treatment of Upper Crossed Syndrome: A Narrative Systematic Review. Healthcare (Basel). 2023 Aug 17;11(16):2328. doi: 10.3390/healthcare11162328. PMID 37628525
- [Background] Ali S, Ahmad S, Jalal Y, Shah B. Effectiveness of Stretching Exercises Versus Muscle Energy Techniques in the Management of Upper Cross Syndrome: JRCRS. 2017; 5 (1): 12-16. Journal Riphah College of Rehabilitation Sciences. 2017;5(1):12-6